CLINICAL TRIAL: NCT03291886
Title: Study of KHK2375 in Subjects With Advanced or Recurrent Breast Cancer
Brief Title: Phase 2 Study of KHK2375 in Subjects With Advanced or Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2375-002
Record Dates: First submitted 2017-09-14; First posted 2017-09-25 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Advanced or Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — entinostat; exemestane

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (exemestane, Entinostat) (Experimental): 5 mg KHK2375 will be administered to subjects once weekly. EXE001 will be administered at a dose of 25 mg once daily orally.
  Pre/perimenopausal female patients also receive luteinizing hormone-releasing hormone (LH-RH) agonist.
  Interventions: Drug: Entinostat; Drug: Exemestane
- Arm B (exemestane, Entinostat(placebo)) (Placebo Comparator): KHK2375 Placebo will be administered to subjects once weekly. EXE001 will be administered at a dose of 25 mg once daily orally.
  Pre/perimenopausal female patients also receive luteinizing hormone-releasing hormone (LH-RH) agonist.
  Interventions: Drug: Entinostat(Placebo); Drug: Exemestane

INTERVENTIONS:
Drug: Entinostat — Given PO
  Other Names: KHK2375; MS-275; SNDX-275
  Arms: Arm A (exemestane, Entinostat)
Drug: Entinostat(Placebo) — Given PO
  Other Names: KHK2375; MS-275; SNDX-275
  Arms: Arm B (exemestane, Entinostat(placebo))
Drug: Exemestane — Given PO
  Other Names: EXE001; Aromasin; FCE-24304

SUMMARY:
The primary objective of this study is to investigate the effect of 5 mg KHK2375 on progression free survival (PFS) when administered orally at weekly intervals in combination with exemestane in a placebo-controlled, double-blind comparative study in subjects with advanced or recurrent hormone receptor-positive breast cancer. The secondary objectives are to investigate the effect of on overall survival (OS) and the antitumor effect and to evaluate the pharmacokinetics and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Personally submitted voluntary written informed consent to participate in the study
2. Age ≥ 20 years at the time of consent
3. Histologically or cytologically confirmed breast cancer positive for estrogen receptor (ER) and/or progesterone receptor (PgR)
4. Human epidermal growth factor 2 (HER2)-negative
5. Stage III/locally advanced or metastatic carcinoma of the breast where local therapy with curative intent is impossible
6. Pre/Peri- and postmenopausal women

   * Postmenopausal status is defined either by:

     1. Age ≥ 55 years and ≥ 1 year of amenorrhea
     2. Age < 55 years and ≥ 1 year of amenorrhea, with blood estradiol (E2) < 20 pg/mL
     3. Age < 55 years with hysterectomy, with ovaries and E2 < 20 pg/mL
   * Surgical menopause with bilateral oophorectomy Pre/perimenopausal women may be enrolled only if they agree to receive an luteinizing hormone-releasing hormone (LH-RH) agonist
7. Eastern Cooperative Oncology Group(ECOG) performance status (PS) of 0 or 1 at enrollment
8. Measurable or nonmeasurable lesions per RECIST version 1.1 criteria
9. Subjects meeting either of the following criteria:

   * History of treatment with a nonsteroidal aromatase inhibitor (AI) for advanced or recurrent breast cancer, and development of progressive disease (PD) after the most recent prior treatment
   * No history of treatment with endocrine therapy for advanced or recurrent breast cancer that has recurred during or within 12 months after postoperative adjuvant therapy with an nonsteroidal AI
10. An adverse event for which a causal relationship to prior treatment cannot be denied (except alopecia) is Grade ≤ 1 in severity or has returned to the baseline level, i.e., the level before the start of the prior treatment
11. The latest laboratory values obtained prior to enrollment must meet all of the following requirements:

    * Hemoglobin concentration: ≥ 9.0 g/dL
    * Platelet count: ≥ 100000/μL
    * Neutrophil count: ≥ 1500/μL
    * Serum creatinine: ≤ 2.0 mg/dL
    * Total bilirubin in serum: < 1.5 × institutional upper limit of normal (≤ 3 mg/dL for subjects with Gilbert's syndrome)
    * Aspartate transaminase(AST) and Alanine transaminase(ALT): ≤ 3.0 × institutional upper limit of normal

Exclusion Criteria:

1. Endocrine therapy (except for LH-RH agonist), treatment with everolimus, treatment with a cyclin-dependent kinase inhibitor, or radiation therapy within 14 days before enrollment

   Subjects with prior treatment with exemestane may be enrolled if they meet either of the following criteria:
   * Start of treatment with exemestane for advanced or recurrent breast cancer within 28 days before enrollment
   * Recurrence-free period >12 months after completion of treatment with exemestane as postoperative adjuvant therapy. For painful bone lesions or impending fractures, radiation therapy may be used concomitantly if there is a measurable or nonmeasurable lesion that is suitable for efficacy evaluation in a region other than the radiation field
2. Two or more prior chemotherapy regimens for advanced or recurrent breast cancer
3. Chemotherapy within 21 days before enrollment
4. Treatment with bisphosphonates or anti-RANKL antibody that is scheduled to be started within 7 days before the first dose of investigational product
5. History of or current central nervous system metastasis, or current leptomeningeal or periosteal disease
6. History of cancer other than breast cancer within 5 years, or concurrent cancer other than breast cancer (except for basal cell carcinoma of skin, squamous cell carcinoma of skin, and intraepithelial carcinoma of uterine cervix).Subjects continuing to receive treatment for cancer other than breast cancer are ineligible for enrollment
7. Ongoing treatment with any other anticancer therapy or investigational product (Except for treatment with exemestane or radiotherapy as described in exclusion criterion 1)
8. Prior treatment with histone deacetylase inhibitor (e.g. valproate, vorinostat)
9. Known allergy to imidazoles, exemestane, or entinostat
10. Any medical or psychiatric condition that could affect compliance with the protocol, ability to give consent, or assessment of anticipated toxicities
11. Uncontrolled complications (e.g., active infections)
12. Positive for either hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus antibody
13. Any other conditions unsuitable for the study in the opinion of the investigator or subinvestigator

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) | Approximately 29 months
  PFS is defined as the number of days from the date of randomization to the date of first documented progressive disease (PD) or the date of death from any cause, whichever comes first (date of first documented PD or death - date of randomization + 1). The date of first documented PD is the date when PD is first documented at overall response assessment or the date when overall response other than complete response (CR) and not evaluable (NE) is documented after first CR. Subjects who receive post-study treatment before the documentation of PD and subjects with no documented PD or death will be censored at the last date they were confirmed to have no PD. Subjects whose overall response from the date of randomization onward is only NE or who have never undergone assessment of antitumor effect, and whose death has not been documented will be censored at the date of randomization.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 50 months
  OS is defined as the number of days from the date of randomization to death from any cause (date of death - date of randomization + 1). Subjects without documented death at the time of data cutoff will be censored at the last date they were confirmed to be alive.
Antitumor effect | Up to 50 months
  The best overall response is defined as the best response recorded from the start of treatment until progression or recurrence according to the categories ordered as CR > partial response(PR) > stable disease (SD) > PD > NE or CR > Non-CR/non-PD > PD > NE. A best overall response of CR or PR will be regarded as objective response. A best overall response of CR, PR, or SD for at least 6 months will be regarded as clinical benefit.

OTHER OUTCOMES:
Plasma concentration of KHK2375 | Day 1 of Cycle 1, Day 15 of Cycle 1 , and Day 1 of Cycle 2 (each cycle is 28 days)
Frequency of subjects with treatment-emergent adverse events | Assessed up to 28 days after study discontinuation

CONTACTS AND LOCATIONS:
Locations (28):
- Japan (28):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Kitakyushu Municipal Medical Center, Kitakyushu, Fukuoka
  - Gunma Cancer Center, Ōta, Gunma
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Tokai University Hospital, Isehara, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Nahanishi Clinic, Naha, Okinawa
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Tokyo Metropolitan Cancer and Infectious Disease Center Komagome Hospital, Bunkyo, Tokyo
  - National Cancer Center Hospital, Chūō, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Toranomon Hospital, Minato, Tokyo
  - Showa University Hospital, Shinagawa, Tokyo
  - Chiba Cancer Center, Chiba
  - Kyushu Cancer Center, Fukuoka
  - Sagara Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka National Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iwata H, Nakamura R, Masuda N, Yamashita T, Yamamoto Y, Kobayashi K, Tsurutani J, Iwasa T, Yonemori K, Tamura K, Aruga T, Tokunaga E, Kaneko K, Lee MJ, Yuno A, Kawabata A, Seike T, Kaneda A, Nishimura Y, Trepel JB, Saji S. Efficacy and exploratory biomarker analysis of entinostat plus exemestane in advanced or recurrent breast cancer: phase II randomized controlled trial. Jpn J Clin Oncol. 2023 Jan 6;53(1):4-15. doi: 10.1093/jjco/hyac166. PMID 36398439